CLINICAL TRIAL: NCT03902639
Title: Comparative Study of the Physiological Effects of High Flow Nasal Cannula and Non-invasive Ventilation in Healthy Volunteers
Brief Title: Examining the Effects of Nasal High Flow Oxygen Therapy Compared to Non-invasive Ventilation in Health Volunteers
Status: Recruiting | Type: Observational
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: REB# 19-006
Record Dates: First submitted 2019-04-02; First posted 2019-04-04 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Healthy Volunteers
Keywords: High flow nasal cannula; Airway pressure; Lung volume; Non-invasive ventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Respiratory failure is characterized by low levels of oxygen and high levels of carbon dioxide in the blood which causes difficulty breathing. The management of patients with respiratory failure aims at improving oxygenation and changing the effort required to breathe. Mechanical ventilation is a life-saving treatment but may be associated with a high mortality rate, prolonged stay in the intensive care unit (ICU), and infection. Oxygenation techniques to avoid mechanical ventilation include standard oxygen therapy, continuous positive pressure (CPAP), and high-flow nasal cannula oxygen therapy (HFNC). CPAP consists of delivering oxygen through a mask. As compared to standard oxygen therapy, CPAP can promote lung recruitment leading to improved oxygenation and the effect in work of breathing in patients with respiratory failure. Conversely, high-flow nasal cannula oxygen therapy (HFNC) delivers oxygen through nasal prongs. Oxygen is heated and humidified and can be delivered at different flows (from 10 - 60 L/min). As compared to standard oxygen therapy, HFNC can promote some lung recruitment leading to mofiy oxygenation and work of breathing. Therefore, the present study will have 2 phases:

Phase 1:Comparison of the physiological effects of different flows of HFNC to CPAP in healthy volunteers. The investigators hypothesized that the physiological effects of HFNC in the nasopharynx are comparable to that of CPAP at 4 cm H2O.

Phase 2: Comparison of the physiological effects of different nasal interfaces of HFNC (Standard cannula vs. Asymmetrical cannula vs. Single-nostril adapted cannula) in healthy volunteers. The investigators hypothesized that the physiological effects of HFNC in the nasopharynx are comparable to that of CPAP at 4 cm H2O. It was hypothesized that asymmetrical which is the cannula that has a higher cross-sectional area generates higher nasal pharyngeal pressure.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers ≥ 18 y-o,
* No evidence of acute or chronic cardiopulmonary disease

Exclusion Criteria:

* Active epistaxis, sinus problem, nasal trauma, or deviated septum that would preclude the nasopharyngeal catheter insertion,
* Pregnancy, clinical evidence of respiratory illness, history of respiratory disease, body mass of over 50 kg/m2, ribcage malformation,
* Cardiac pace maker or implantable cardioverter-defibrillator according to EIT manufacturer,
* Allergy to topical lidocaine,
* Claustrophobia that would preclude the use of CPAP or HFNC.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers responding to advertisement posted through the St. Michael's Hospital Communications board.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2019-04-10 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
End expiratory nasopharyngeal pressure (NP) | 5 minutes
  The primary endpoint is to compare the end expiratory nasopharyngeal pressure (NP) under 60 L/min of high flow nasal cannula (HFNC) to continuous positive airway pressure (CPAP 4 cmH2O).This will be assessed using a nasopharyngeal catheter.
End expiratory nasopharyngeal pressure (NP) | 5min
  The primary endpoint is to compare the end expiratory nasopharyngeal pressure (NP) of high flow nasal cannula (HFNC) among the 3 different nasal cannulas (Symmetrical, Asymmetrical, Single-nostril adapted).

SECONDARY OUTCOMES:
Change in physiologic variables of airway pressure at different flows of HFNC (20, 40, and 60 L/min) and CPAP (4 cmH20). In the phase#2; HFNC 2, and 50 L/min. | 5 minutes
  One of the secondary endpoints is to compare variables of airway pressure at different flows of HFNC to CPAP. The investigators will measure the end expiratory NP, mean NP, mean peak inspiratory pressure, mean peak expiratory pressure, delta inspiratory pressure and delta expiratory pressure.
  Each of these variables will be measured for 1 minute using a nasopharyngeal catheter. Furthermore, at each flow of HFNC, the investigators will ask the patient to breathe with their mouth open and mouth closed.
Change in end-expiratory lung impedance | 5 minnutes
  The other secondary endpoint is to compare the change in ventilation distribution and end-expiratory lung impedance at different flows of HFNC and CPAP (Different nasal cannulas in the 2nd phase). These variables will be measured using electrical impedance tomography (EIT) by placing a band around the chest of each participant.
Dead-space washout in the upper airways | 5 minutes
  Assess whether the transcutaneous CO2 is modified by HFNC, while comparing 3 different nasal cannulas (Symmetrical, Asymmetrical, Single-nostril adapted).

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Brochard, MD, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No